CLINICAL TRIAL: NCT07168993
Title: Detection of Early-Stage Lung Cancer in Sputum Using Flow Cytometry and an Automated Analysis Pipeline
Brief Title: Evaluate the Clinical Performance of the Flow Cytometry - FlowPath Lung Test as a Sensitive and Specific Non-invasive Diagnostic of Sputum Samples to Identify/Detect the Presence of Lung Cancer in High-risk Individuals Who Have Existing Lung Nodules, >6 to <30 mm in Diameter, Determined by LDCT.
Acronym: BA-004
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: bioAffinity Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BA-004
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: Lung Cancer; Diagnostic Test; Sputum Assay
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Diagnostic testing of sputum sample provided by subject
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Other: Standard medical treatment — Standard of care follow up per institution
  Other Names: Standard of care follow up per institution
Other: Standard medical treatment — SOC per institution
  Other Names: Follow up SOC

SUMMARY:
Evaluate FlowPath Lung Diagnostic Test of Sputum Samples to Detect the Presence of Lung Cancer in High-risk Individuals Who Have Existing Lung Nodules, >6 to <30 mm in Diameter, Determined by LDCT.

DETAILED DESCRIPTION:
Evaluate the Clinical Performance of the Flow Cytometry - FlowPath Lung Test as a Sensitive and Specific Non-invasive Diagnostic of Sputum Samples to Identify/Detect the Presence of Lung Cancer in High-risk Individuals Who Have Existing Lung Nodules, >6 to <30 mm in Diameter, Determined by LDCT.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to give signed informed consent and comply with study requirements.
2. Is high risk for getting lung cancer:

   1. ≥50 - 80 years of age.
   2. current smoker with smoking history of at least 20 pack-years or current non-smoker with smoking history of at least 20 pack-years who quit smoking within the past 15 years.
3. Has a >6 to <30 mm diameter lung nodule (found by lung cancer screening or found incidentally by CT scan) as determined by CT and is willing to provide a sputum sample for FlowPath Lung test within 6 weeks of the prestudy baseline CT scan.

3a) Nodule is either new, increasing, or stable for ≤ 6 months. 3b) In cases where a person has multiple nodules as determined by CT scan, the subject's most suspicious nodule is >6 to <30 mm in diameter.

4) Is willing to provide contact information to the study PI or the treating physician(s) who can release required medical information related to SOC follow-up.

Exclusion Criteria:

1. Is unable to cough with sufficient exertion to produce a sputum sample (e.g., due to severe obstructive lung disease).
2. The dominant nodule is ground glass or part solid as determined by CT scan.
3. Has 5 or more nodules sized >4 mm.
4. The nodule sized >6 to <30 mm in diameter is a distal (subsegmental) endobronchial nodule or a perifissural nodule.
5. Is immunosuppressed.
6. Has rheumatoid arthritis.
7. Had lung cancer diagnosis in the past 5 years or any other cancer (other than non-melanoma skin cancer) in the past 2 years. A subject on long-term medications used for prevention of cancer, such as Tamoxifen for breast cancer, is not excluded.
8. Has angina with minimal exertion.
9. Is currently pregnant or planning on becoming pregnant during this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2063 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate FlowPath Lung Test Detection of Early-Stage Lung Cancer in Sputum | From Baseline Sputum Sample provided by subject through 24 months follow up period.
  Evaluate the clinical performance (positive percent agreement [PPA/sensitivity] and negative percent agreement [NPA/specificity]) of the FlowPath Lung test in predicting lung cancer from the sputum of high-risk individuals with lung nodules

IPD SHARING:
Plan to Share IPD: Undecided